CLINICAL TRIAL: NCT05102006
Title: A Multicenter Phase Ib/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of LBL-007 in Combination With Toripalimab in the Treatment of Advanced Malignancies
Brief Title: A Phase Ib/II Clinical Study of LBL-007 in Combination With Toripalimab in Treatment of Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LBL-007-CN-003
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Advanced Malignant Tumors
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LBL-007&Toripalimab (Experimental): LBL-007 Injection; dose A or dose B; Q3W
  Toripalimab Injection; dose C; Q3W
  Interventions: Drug: LBL-007 Injection; Drug: Toripalimab Injection

INTERVENTIONS:
Drug: LBL-007 Injection — LBL-007 Injection; dose A or dose B; Q3W
  Other Names: LBL-007
Drug: Toripalimab Injection — Toripalimab Injection; dose C; Q3W
  Other Names: Toripalimab

SUMMARY:
This is a single-arm, open-label, multicenter Phase Ib/II clinical study to evaluate the safety, tolerability, PK characteristics, immunogenicity and efficacy of LBL-007 in combination with Toripalimab in Treatment of Advanced Malignant Tumors.

DETAILED DESCRIPTION:
This trial is divided into combination dose escalation phase (Phase Ib) and combination dose expansion phase (Phase II), as follows:

1. In the Phase Ib study, patients with advanced neoplasm malignant who have no standard treatment or have treatment failure of standard treatment or are not suitable for standard treatment at present stage are planned to be enrolled,including patients with advanced neoplasm malignant who have not been treated with anti-PD- (L) 1 antibody or have progressed or not tolerated after treatment with anti-PD- (L) 1 antibody.LBL-007 is administered once every 3 weeks (Q3W),intravenous infusion.The dosing regimen of toripalimab in combination was once every 3 weeks (Q3W),Intravenous infusion.
2. According to the LBL-007 global research and development data and the safety, tolerability and PK data of the phase Ib clinical study, the recommended dose of phase II clinical study (RP2D) was obtained for the expansion of target indications.This study is designed to enroll patients with advanced neoplasm malignant, including patients who have not been treated with anti-PD- (L) 1 antibody or patients who have progressed or intolerant after treatment with anti-PD- (L) 1 antibody.Subjects need to undergo relevant examinations or observations during the screening period,and subjects who meet the screening requirements will enter the treatment period.
3. Biological samples will be collected from subjects in Phase Ib/II for relevant testing in this trial.Phase Ib is expected to enroll approximately 9-12 subjects.Phase II is expected to enroll approximately 200 subjects.The number of subjects to be enrolled was determined by actual conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen and visit schedule, voluntarily enroll in the study, and sign the written informed consent form.
2. Age ≥ 18 and ≤ 75 years at the time of signing the informed consent, regardless of gender.
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1.
4. The expected survival time is at least 12 weeks.
5. Males with fertility and females of childbearing age are willing to take highly effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug (including abstinence, intrauterine device, various hormonal contraception, correct use of contraception Sets，etc）;Women of childbearing age include pre-menopausal women and women within 2 years after menopause. Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.

Exclusion Criteria:

1. Have received other unmarketed clinical investigational drugs or treatments within 4 weeks prior to the first dose of study drug.
2. Use of immunomodulatory drugs within 14 days before the first use of the study drug, including but not limited to thymopeptide, interleukin-2, interferon, etc..
3. Patients with active infection and currently requiring intravenous anti-infective therapy.
4. Patients with clinically uncontrollable pleural effusion, pericardial effusion or ascites, and those requiring repeated drainage or medical intervention.
5. The patient has a Medical history of immunodeficiency, including HIV antibody positive.
6. Active hepatitis B or active hepatitis C.
7. Women during pregnancy or lactation.
8. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour) or Lugano 2014 (lymphoma),Proportion of subjects achieving complete response (CR) or partial response (PR).It was used to evaluate the efficacy in Phase II
Dose-limiting toxicities（DLT） | During the first Cycles(each cycle is 21 days)
  DLT describes side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.DLT is defined as toxicity (possible adverse events related to LBL-007) during the DLT observation period (3 weeks after the first dose).It was used to evaluate the safety in Phase Ib.
Maximum tolerated dose (MTD) | During the first Cycles(each cycle is 21 days)
  MTD is defined as the hightest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycles. It was used to evaluate the tolerability in Phase Ib .

SECONDARY OUTCOMES:
Number of subjcects with adverse events and serious adverse events | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Adverse event (AE) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.The safety profile of LBL-007 and Toripalimab will be assessed by monitoring the Adverse event (AE).
Disease Control Rate(DCR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR, PR, iCR, iPR and stable disease (SD) after treatment.
Duration of Response(DOR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  DOR is defined as the duration from earliest date of disease response (CR、PR 、iCR or iPR) until earliest date of disease progression or death from any cause(if occurring sooner than progression).
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (30+7 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.Immunogenicity refers to the performance that can elicit an immune response.

CONTACTS AND LOCATIONS:
Overall Officials: li zhang, Principal Investigator — Sun Yat-sen University
Locations (14):
- China (14):
  - The first affiliated hospital of bengbu medical University, Bengbu, Anhui
  - Chongqing University Three gorges Hospital, Chongqing, Chongqing Municipality
  - The 900 Hospital of the Joint Service Support Force of the People's Liberation Army of China, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First People's Hospital of Yu Lin, Yulin, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Changzhou Cancer Hospital, Changzhou, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No